CLINICAL TRIAL: NCT05876000
Title: Prospective Multi-Center Single-Arm Study for Evaluating the Corheart 6 Left Ventricular Assist System
Brief Title: Corheart 6 LVAS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_EU_LVAS
Record Dates: First submitted 2023-04-24; First posted 2023-05-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Refractory Heart Failure
Keywords: Advanced Heart Failure; Left Ventricular Assist System; Mechanical Circulatory Support
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corheart 6 LVAS (Experimental): The Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) to be used on patients with advanced left ventricular heart failure.
  Interventions: Device: Corheart 6 Left Ventricular Assist System

INTERVENTIONS:
Device: Corheart 6 Left Ventricular Assist System — Implantation of left ventricular assist device for mechanical circulatory support

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the Corheart 6 LVAS when used for the treatment of advanced left ventricular heart failure in a European population at 6 months post-implantation.

The secondary objective is to assess the long-term safety and effectiveness of Corheart 6 LVAS treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years and ≤ 75 years
* 2. The patient has signed an Informed Consent Form
* 3. Body Surface Area (BSA) ≥ 1.2 m^2
* 4. New York Heart Association (NYHA) Class IV
* 5. Left Ventricular Ejection Fraction (LVEF) ≤ 25%
* 6. Despite the optimal medical management based on current guidelines, the patient must also meet one or more of the following:
* a. Unable to exercise for HF,
* or
* if able to perform cardiopulmonary testing, with peak VO2 <12 mL/kg/min and/or < 50% predicted value;
* b. Progressive end-organ dysfunction (worsening renal and/or hepatic function, type II pulmonary hypertension, cardiac cachexia) due to reduced perfusion and not to inadequately low ventricular filling pressure (PCWP > 20 mmHg and SBP < 90 mmHg or CI < 2.0 L/min/m2).
* c. Impella or IABP assisted;
* d. Inotrope dependent/unable to wean from inotropes.

Exclusion Criteria:

* 1. Heart failure who can be treated with other therapy options (e.g. CRT, CRT-D, etc.)
* 2. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the patients' health status.
* 3. Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia type II.
* 4. Platelet count < 100,000 x 10^3/L (< 100,000/ml).
* 5. Psychiatric disease/ disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and ventricular assist system management.
* 6. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator.
* 7. Presence of an active, uncontrolled infection.
* 8. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:
* a. Total bilirubin > 51.3 μmol/L (3.0 mg/dl), ischemic hepatitis, or biopsy proven liver cirrhosis, or clinically Child-Pugh B and C score.
* b. History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, or FEV1 < 50% predicted.
* c. Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention.
* d. History of stroke within 180 days prior to enrollment, or a history of cerebrovascular disease with symptomatic (> 70%) carotid artery stenosis
* e. Serum creatinine ≥ 265 μmol/L (3.0mg/dl) or requiring dialysis.
* f. Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration.
* 9. Etiology of heart failure (HF) due to or associated with uncorrected thyroid disease, obstructive/ restrictive cardiomyopathy, pericardial disease, amyloidosis or giant cell myocarditis.
* 10. Uncorrected moderate to severe aortic insufficiency without plans for correction during pump implant.
* 11. History of confirmed, untreated abdominal aortic aneurysm (AAA) or thoracic aortic aneurysm (TAA) > 5 cm in diameter.
* 12. Uncontrollable ventricular tachyarrythmias/ ventricular fibrillation (VF).
* 13. STEMI <2 weeks before planned implantation.
* 14. Right ventricular failure as defined by one or more of the following:
* a. severe depressed RV function in echocardiography
* b. TAPSE < 1.0 cm
* c. CVP/PCWP ratio > 0.63
* 15. Planned Bi-VAD support prior to enrollment.
* 16. Cardiac arrest with a history of resuscitation 1-month before inclusion, without full restoration of cognitive function.
* 17. History of any organ transplant.
* 18. Pre albumin < 150 mg/L, or Albumin < 30g/L (3 g/dL).
* 19. Any condition other than HF that could limit survival to less than 24 months.
* 20. Positive pregnancy test if of childbearing potential.
* 21. Lactating mothers.
* 22. Participation in any other clinical investigation that is likely to confound study results or affect the study.
* 23. Patients who have been placed in an institution by court order or by order of the authorities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of surivival | Up to 6 months post-implantation
  At 6 months post-implantation, composite of survival to transplant, recovery, LVAS support free of disabling stroke (Modified Rankin Score > 3), or re-operation to replace the pump due to pump failure.

SECONDARY OUTCOMES:
Survival | Year 1, Year 2, Year 3, Year 4, Year 5
  Overall survival of patients
Composite of surivival | Year 1, Year 2, Year 5
  Composite of survival to transplant, recovery, LVAS support free of disabling stroke (Modified Rankin Score > 3), or re-operation to replace the pump due to pump failure.
Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, Month 3, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  Scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.
Quality of Life as measured by the EuroQoL-5D-5L (EQ-5D-5L) | Baseline, Month 3, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  The scores from the 5 dimensions are summed for the total score which ranges from 5 to 25 with higher scores indicating more problems and a worse quality of life.
Functional status as measured by the Six Minute Walk Test (6MWT) | Baseline, Month 3, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  The more meters a patient can walk over baseline indicates improvement in functional status.
Functional status as measured by the New York Heart Association (NYHA) Classification | Baseline, Month 3, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  NYHA class categorizes patients by the severity of their heart failure symptoms. As the class increases, the degree of symptoms is more severe indicating worse functional status.
Adverse Events | As they occurred, from Baseline to Year 5
  Frequency and incidence of all anticipated Adverse Event.

CONTACTS AND LOCATIONS:
Overall Officials: Evgenij V Potapov, Principal Investigator — German Heart Institute
Locations (11):
- Austria (2):
  - Universitätsklinikum Graz, Graz
  - Universitätskliniken der MedUni Wien, Vienna
- Germany (7):
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Deutsches Herzzentrum der Charité, Berlin
  - Klinikum Links der Weser, Bremen
  - Universitätsklinikum Hamburg, Hamburg
  - Universitätsklinikums Heidelberg, Heidelberg
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Würzburg, Würzburg
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: Undecided
At this moment the IPD is not yet available for access and will be updated when it is ready.